CLINICAL TRIAL: NCT03370666
Title: High Flow Nasal Therapy Versus Noninvasive Ventilation in Mild to Moderate Acute Hypercapnic Respiratory Failure: A Non-inferiority Randomized Trial
Brief Title: High Flow Nasal Therapy Versus Noninvasive Ventilation in COPD Exacerbation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone Palermo (Other)
Collaborators: Azienda Ospedaliera Universitaria Mater Domini, Catanzaro (Other)
Responsible Party: Principal Investigator, Andrea Cortegiani, MD, Principal Investigator, Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone Palermo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07/17
Record Dates: First submitted 2017-11-29; First posted 2017-12-12 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: COPD Exacerbation

STUDY DESIGN:
Intervention Model Description: Non-inferiority
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFNT (Experimental): HFNT performed with any available device. The flow will be initially set at 60 liters per minute and temperature at 37° C. The target will be an oxygen saturation (SpO2) of 88-92%. In case of patient not tolerating these settings, flow and temperature will be titrated to the maximum tolerated level.
  Interventions: Other: HFNT
- NIV (Active Comparator): NIV must be delivered by full or oronasal mask with any available ventilator. The ventilator settings will be decided according to the usual practice: maximal tolerated inspiratory pressure to obtain a measured or estimated expired tidal volume of 6-8 mL·kg-1 of body weight and a positive end expiratory pressure (PEEP) between 3 and 5 cmH2O. An interface rotational strategy will be allowed among only different types of masks.
  Interventions: Other: NIV

INTERVENTIONS:
Other: HFNT — High flow nasal therapy
  Arms: HFNT
Other: NIV — Noninvasive ventilation
  Arms: NIV

SUMMARY:
Randomized multicenter non-inferiority trial comparing High flow nasal therapy (HFNT) versus Noninvasive ventilation (NIV) in patients with chronic obstructive pulmonary disease (COPD) and acute hypercapnic respiratory failure.

DETAILED DESCRIPTION:
The interventions will be delivered in Emergency Departments or Intensive Care Units.

The intervention under investigation will be High flow nasal therapy. Investigators will deliver HFNT to enrolled patients using any available device able to produce it. The flow will be initially set at 60 liters per minute and temperature at 37° C. The target will be an oxygen saturation (SpO2) of 88-92%. In case of patient not tolerating these settings, flow and temperature will be titrated to the maximum tolerated level. The intervention will last until one of the following conditions: 1) physician in charge decide to interrupt HFNT and start NIV because the patient shows signs of persisting worsening respiratory failure; 2) physician in charge decide to interrupt HFNT and perform endotracheal intubation and invasive mechanical ventilation because patient shows one or more of these conditions: respiratory arrest, respiratory pauses with loss of consciousness, psychomotor agitation making nursing care impossible, heart rate < 50 with loss of alertness, hemodynamic instability with systolic arterial blood pressure <70 mmHg, development of conditions requiring intubation either to protect the airway or to manage copious tracheal secretions, inability to tolerate the devices; 3) clinical improvement defined as all these conditions: normal mental status, hemodynamic stability, respiratory rate below 25 per minute, absence of activation of accessory respiratory muscles and paradoxical abdominal motion, no dyspnea arterial pH > 7.35, Arterial partial pressure of carbon dioxide (PaCO2) < 70 mmHg and Arterial partial pressure of oxygen (PaO2) > 55 mmHg with an inspired oxygen fraction (FiO2) < 0.35.

In case of temporary interruption of the intervention for any cause, patients should receive oxygen supplementation with Venturi mask with a target of SpO2 88-92%.The comparator will be non invasive ventilation (NIV). NIV must be delivered by full or oronasal mask. The ventilator settings will be decided according to the usual practice: maximal tolerated inspiratory pressure to obtain a measured or estimated expired tidal volume of 6-8 mL·kg-1 of body weight and a positive end expiratory pressure (PEEP) between 3 and 5 cmH2O. An interface rotational strategy will be allowed among only different types of masks.

The intervention will last until one of the following conditions: 1) physician in charge decide to interrupt NIV and perform endotracheal intubation and invasive mechanical ventilation because patient shows one or more of these conditions: respiratory arrest, respiratory pauses with loss of consciousness, psychomotor agitation making nursing care impossible, heart rate < 50 with loss of alertness, hemodynamic instability with systolic arterial blood pressure <70 mmHg, development of conditions requiring intubation either to protect the airway or to manage copious tracheal secretions, inability to tolerate the devices; 2) clinical improvement defined as all these conditions: normal mental status, hemodynamic stability, respiratory rate below 25 per minute, absence of activation of accessory respiratory muscles and paradoxical abdominal motion, no dyspnoea arterial pH > 7.35, Arterial partial pressure of carbon dioxide (PaCO2) < 70 mmHg and Arterial partial pressure of oxygen (PaO2) > 55 mmHg with an inspired oxygen fraction (FiO2) < 0.35.

In case of temporary interruption of NIV for any cause, patients should receive oxygen supplementation with Venturi mask with a target of SpO2 88-92%.

ELIGIBILITY:
Inclusion Criteria:

* Presence of chronic obstructive pulmonary disease (COPD) and acute hypercapnic respiratory failure;
* 7.25 < pH < 7.35;
* Arterial Partial pressure of carbon dioxide (PaCO2) equal or greater than 55 mmHg;
* Age > 18 years/old

Exclusion Criteria:

* Invasive mechanical ventilation in the last 60 days
* Use of any form of noninvasive ventilation or high flow oxygen through nasal cannula (HFNT) prior to study enrollment after the onset of acute hypercapnic respiratory failure (AHRF);
* Noninvasive home care ventilation;
* Unstable clinical condition (need for vasopressors for >24 h, acute coronary syndrome or life-threatening arrhythmias);
* Refusal of treatment;
* Agitation (RASS >= +2) or non-cooperation (Kelly Matthay >=5);
* Failure of more than two organs;
* Cardiac arrest;
* Respiratory arrest requiring tracheal intubation;
* Recent trauma or burns of the neck and face;
* Pregnancy;
* Refusal of consent;
* Inclusion in other research protocols.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
Arterial partial pressure of carbon dioxide (PaCO2) | 2 hours after randomization

SECONDARY OUTCOMES:
Dyspnea evaluated with Borg dyspnea scale | 2 and 6 hours after randomization
  Borg dyspnea scale: this is a 12-point validated scale that rates patient's difficulty in breathing. It starts at number 0 where breathing causes no difficulty at all and progresses through number 10 where breathing difficulty is maximal
Arterial partial pressure of carbon dioxide (PaCO2) | 6 hours after randomization

OTHER OUTCOMES:
Respiratory rate | 2 and 6 hours after randomization
Discontinuation of the interventions | At 6 hours after randomization
  The inability of the patient to continue the treatment while there was still an indication for ventilatory support
Overall discomfort related to the interface | At 6 hours after randomization
Presence of side effects | At 6 hours after randomization
  I.e., complaining for noise or too high temperature of flow, claustrophobia, gastric distension, vomiting, sweating, tightness
Rate of treatment failure | At 6 hours after randomization
  defined as the presence of one or more of the following: arterial partial pressure of carbon dioxide (PaCO2) reduction, no change or reduction < 10 mmHg from baseline, worsening or no improvement in dyspnoea, respiratory rate > 30 breaths per minute, use of accessory respiratory muscles or paradoxical abdominal movement
Rate of endotracheal intubation | At 6 hours after randomization
  Number of patients requiring endotracheal intubation

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Navalesi, MD, Study Director — Azienda Ospedaliera Universitaria Mater Domini, Catanzaro
Locations (10):
- Italy (10):
  - Ospedale S. Donato, Arezzo
  - Ospedale Sant'Orsola Malpighi. Università Alma Mater, Bologna
  - A.O.U. Policlinico-Vittorio Emanuele, Università degli Studi di Catania, Catania
  - Azienda Ospedaliera Universitaria Mater Domini, Catanzaro
  - University Hospital of Modena, Pneumology Unit and Center for Rare Lung Diseases, Department of Medical and Surgical Sciences, University of Modena and Reggio Emilia, Modena
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone. Università degli Studi di Palermo, Palermo
  - IRCCS Maugeri, Pavia
  - Azienda Ospedaliera di Perugia, Perugia
  - Ospedale Molinette, Torino
  - Azienda Sanitaria Universitaria Integrata di Udine, Udine

REFERENCES:
- [Derived] Cortegiani A, Longhini F, Madotto F, Groff P, Scala R, Crimi C, Carlucci A, Bruni A, Garofalo E, Raineri SM, Tonelli R, Comellini V, Lupia E, Vetrugno L, Clini E, Giarratano A, Nava S, Navalesi P, Gregoretti C; H. F.-AECOPD study investigators. High flow nasal therapy versus noninvasive ventilation as initial ventilatory strategy in COPD exacerbation: a multicenter non-inferiority randomized trial. Crit Care. 2020 Dec 14;24(1):692. doi: 10.1186/s13054-020-03409-0. PMID 33317579
- [Derived] Cortegiani A, Longhini F, Carlucci A, Scala R, Groff P, Bruni A, Garofalo E, Taliani MR, Maccari U, Vetrugno L, Lupia E, Misseri G, Comellini V, Giarratano A, Nava S, Navalesi P, Gregoretti C. High-flow nasal therapy versus noninvasive ventilation in COPD patients with mild-to-moderate hypercapnic acute respiratory failure: study protocol for a noninferiority randomized clinical trial. Trials. 2019 Jul 22;20(1):450. doi: 10.1186/s13063-019-3514-1. PMID 31331372